CLINICAL TRIAL: NCT04919525
Title: Remote Gamified Sensory Perceptual Training for Patients With Fibromyalgia: a Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Laura Tabacof, Postdoctoral Fellow, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB-20-01292
Record Dates: First submitted 2021-05-05; First posted 2021-06-09 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Fibromyalgia
Keywords: Gamified; Somatosensory; Temporal discrimination; Cognitive training; Chronic Pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TrainPain Intervention (Experimental): Daily TrainPain protocol - gamified sensory perceptual training
  Interventions: Device: TrainPain

INTERVENTIONS:
Device: TrainPain — Participants will use gamified sensory perceptual training technology once daily for 28 days. This will involve participants completing a 15 minute sensory training session using the provided technology and viewing a 5 minute web based pain management lesson; additionally, participants will receive daily text messages. The device used in this study has two components. The first is a video game that can be downloaded onto any smartphone device. The second component is two vibrational devices that can be attached to the arms, legs, upper back, and lower back.

SUMMARY:
The purpose of this study is to determine the feasibility of gamified sensory perceptual training in people with fibromyalgia. The primary aim is to determine the feasibility of at-home somatosensorial training for people with fibromyalgia. The researchers are determining the feasibility of using this device to decrease chronic neuropathic pain in people with fibromyalgia. The secondary aim is to survey participants' subjective report of clinical change after this program.

DETAILED DESCRIPTION:
Fibromyalgia is a pain syndrome characterized by central sensitization, and hypersensitivity to nociceptive stimuli. In people with fibromyalgia, objective measures of sensory perception are often impaired. For example, somatosensory temporal discrimination thresholds are elevated, and this correlates with increased widespread pain and severity of other symptoms including fatigue, sleep quality, cognitive symptoms, somatic symptoms and decreased functional status. Sensory-Cognitive training may reduce symptoms by improving attentional modulation of somatosensory signals, improving precision of sensory discrimination, and altering affective processing of somatosensation. The objective of this study is to evaluate the feasibility of the TrainPain program as a somatosensory therapy for people with fibromyalgia.. This study plans to enroll 30 participants between the ages of 18 and 65 who are diagnosed with fibromyalgia and have been experiencing chronic pain with an NRS rating of 4/10 for at least 3 months. All participants who agree to participate in this study will answer a set of baseline questionnaires (PEG, FAS) about their symptoms at the time of inclusion. Participants will also receive the device, and view a demonstration of how to use the technology. The technology consists of two components; (1) an application downloaded to the participants' smartphone and (2) two vibrational devices to be placed on the body of the participant, connected to the application via bluetooth. Participants will use this technology once daily for 28 days. Participants will complete a 15 minute sensory training session using the provided technology; additionally, participants will receive daily text messages to promote pain self-management, and program adherence. Participants will also complete the PEG questionnaire once weekly. After 28 days study team members will conduct a virtual follow-up visit. In that visit, participants will complete the same questionnaires as at baseline (PEG, FAS), as well as a question on their perception of clinical change (PGIC). Participants will also be asked to complete the system usability scale and provide a net promoter score. Finally, participants will complete a subjective feedback questionnaire where they will rate whether participating in this program was time well spent and enjoyable. The primary aim is to determine the feasibility of at-home somatosensorial training for people with fibromyalgia. The secondary aim is to survey participants' subjective report of clinical change after this.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 65 at consent
* Chronic pain ( at least 3 months)
* Minimum average pain of 4 in the NRS

Exclusion Criteria:

* Not able to comprehend English written language
* Chronic skin disease or topical allergies that would be worsened by the use of sensor tape
* Severe psychiatric disorder (Patient Health Questionnaire)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Retention rates | 5 weeks
  Retention rates to assess the feasibility of at-home somatosensorial training technology for people with fibromyalgia
Adherence rates | 5 weeks
  Adherence rates to the assess feasibility of at-home somatosensorial training technology for people with fibromyalgia
The System Usability Score | 5 weeks
  Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking.
The Net Promoter Score | 5 weeks
  The Net Promoter Score is an index ranging from 0-10 that measures the willingness of customers to recommend a company's products or services to others as a measure of opinion on the feasibility on using the device. Higher score indicates higher recommendation.
The Subjective Feedback Questionnaire | 5 weeks
  The Subjective Feedback Questionnaire asks participants to rate the acceptability, enjoyment, and perceived usefulness (0-10) of the program as a measure of opinion on the feasibility on using the device. Higher score indicates higher enjoyment. There are also 12 subjective yes/no questions asking participants to report their opinions of the program and its affect on their pain and quality of life. Finally, there are two open-ended questions that give participants the opportunity to provide feedback on the program.

SECONDARY OUTCOMES:
Change The Pain, Enjoyment of Life and General Activity (PEG) Scale | Baseline and 5 weeks
  The Pain, Enjoyment of Life and General Activity (PEG) Scale consists of 3 separate numerical scales. Each scale has ratings ranging from 0-10. The PEG scale is scored by averaging the three numbers. Full scale from 0-10, higher score indicates worse pain, and pain interference. Change in score at 5 weeks compared to baseline.
Change Patient Global Impression of Change (PGIC) | Baseline and 5 weeks
  The Patient's Global Impression of Change (PGIC) Full score from -3 to 3, with higher score indicating more improvement. Change in score at 5 weeks compared to baseline.
Pain Catastrophizing Scale (PCS) | Baseline and 5 weeks
  The PCS contains 13 questions. The full score ranges from 0 to 39 where a higher score correlates with more extreme pain catastrophization.
Change in Fibromyalgia Assessment Scale (FAS) | Baseline and 5 weeks
  Fibromyalgia Assessment Scale (FAS) is a short and easy to complete self-administered index combining a set of questions relating to non-articular pain (SAPS range 0 to 10), fatigue (range 0 to 10), and the quality of sleep (range 0 to 10) that provides a single composite measure of disease activity ranging from 0 to 10. higher score indicates poorer health outcomes. Change in score at 5 weeks compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Tabacof, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No